CLINICAL TRIAL: NCT04630574
Title: Characterization and Quantification of Motor Speech Disorders in Huntington's Disease: Identification of Acoustic Markers
Acronym: TPMH
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/67
Record Dates: First submitted 2020-11-01; First posted 2020-11-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; Dysarthria; Motor speech performance; Acoustic markers
MeSH Terms: conditions — Huntington Disease; Dysarthria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Huntington's disease: Each patient is seen in the framework of his annual follow-up consultation, for an evaluation of his speech with the computerized tool MonPaGe.
  Interventions: Other: Speech evaluation with the clinical evaluation of dysarthria; Other: complete assessment of the MonPaGe computerized protocol

INTERVENTIONS:
Other: Speech evaluation with the clinical evaluation of dysarthria — A first speech evaluation with the clinical evaluation of dysarthria during 30 minutes is proposed to exclude very severe dysarthria.
Other: complete assessment of the MonPaGe computerized protocol — The application records directly and anonymously stores speech productions made by the patient.

SUMMARY:
The study proposes to identify deviant speech dimensions in patients with HD at presymptomatic and declared stages of the disease, compared to healthy subjects, using the computerized MonPaGe speech protocol. This tool is based on a multidimensional and quantified assessment of voice and speech, by a set of targeted acoustic and perceptual criteria.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a neurodegenerative disorder of the central nervous system, of genetic etiology. It manifests itself in motor, cognitive and psychiatric disorders, which progressively worsen until the patient is grabbed. Motor speech performance disorders are present from the early stage of the disease. These difficulties, which progressively worsen until the end of the patient's life, lead to a communication disorder and constitute a major handicap with social withdrawal, loss of self-esteem and isolation, which are always very painfully experienced by patients and their entourage. Dysarthria in the HD has been very little studied, which makes its speech therapy uncodified. According to the most widely used classification by speech therapists and neurologists, the Darley classification (1975), the speech disorders observed in the HD are included in the heterogeneous group of hyperkinetic dysarthria, whose contours and properties are ill-defined. In this context, a more precise knowledge of speech disorders in the HD appears necessary to identify and characterize the different types of dysarthria and the dysfunctions associated with each level of production (respiration, phonation, resonance, articulation, prosody) and thus improve speech language therapy.

The investigators propose to use an acoustic evaluation to support the perceptual evaluation, available in the MonPaGe protocol, to describe the fine characteristics of the speech disorders in the HD and to define objective markers of dysarthria in this disease for francophone patients.

Each patient is seen in the framework of his annual follow-up consultation in the Competence Center mdH of Bordeaux University Hospital or in the Reference Center mdH of the hospital Henri Mondor of Créteil, for an evaluation of his speech with the computerized tool MonPaGe. A first speech evaluation with the BECD (Auzou, 2006) during 30 minutes is proposed to exclude very severe dysarthria. At the end of this rapid test subtest, the subjects who obtain a perceptive score <16 are offered the complete assesment of the MonPaGe computerized protocol (30 minutes).The application records directly and anonymously stores speech productions made by the patient.The productions are transmitted to the Phonetics and Phonology Laboratory of Paris (UMR 7018 CNRS / Sorbonne Nouvelle), via a secure large data exchange server and are subject to a perceptual and acoustic evaluation a posteriori.

ELIGIBILITY:
Inclusion Criteria:

* major patients
* francophone patients
* Huntington's disease carriers confirmed by molecular biological analysis
* carriers of pre-symptomatic Huntington's disease: Total Motor Score of the Unified Huntington's Disease Rating Scale <5
* carriers of Huntington's disease at a declared stage: Total Motor Score of the Unified Huntington's Disease Rating Scale ≥ 5
* followed in the Competence Center Huntington's disease Bordeaux Hospital or in the Reference Center Huntington's disease Henri Mondor Hospital of Créteil
* affiliates or beneficiaries of a social security scheme
* Finally, a free, informed and express consent of the patient must be collected.

Exclusion Criteria:

* Huntington's disease patients with severe dysarthria (BECD score> 16), acoustic analysis not being possible on unintelligible speech
* patients placed under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Huntington's disease at presymptomatic and declared stages of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Determination of the intelligibility score. | Day 1
  Defined as the number of words correctly recognized by the evaluator (score out of 15).
Determination of the maximum phonation time. | Day 1
  Expressed in milliseconds.
Determination of the phonation characteristics. | Day 1
  Described as the mean and standard deviation of fundamental frequency (in Hz),
Determination of the intensity modulation capacities. | Day 1
  Based on a scale of 0 to 4.
Determination of the Coarticulation. | Day 1
  Expressed in Hz. Extracted from the spectral properties of the acoustic signal of certain words.
Determination of the prosody. | Day 1
  assessed on a scale 0 to 4 on particular sentences.
Determination of the diadocokinesies, | Day 1
  assessed on two scales: precision (0 to 4) and control (0 to 4).
Determination of the articulation rate. | Day 1
  expressed in syllabs per second.

SECONDARY OUTCOMES:
Determination of the Huntington's disease stage. | Day 1
  The Huntington's disease stage will be determined based on the Total Functional Capacity (TFC) and the Total Motor Score (TMS) scales of the Unified Huntington's Disease Rating Scale:
  * pre-symptomatic stage: TFC = 13 / TMS <5
  * light stage: TFC ≥11 / TMS 5 to 20
  * moderate stage: TFC = 7 to 10 / TMS: 20 to 40
Determination of the clinical motor forms of the Huntington's disease. | Day 1
  The clinical motor forms of Huntington disease will be determined by the motor UHDRS scale (Total Motor Score), which evaluates oculomotricity, skill and manual planning, bradykinesia, dystonia and rigidity, chorea and walking, balance, lingual protrusion and dysarthria.
Determination of the level of cognitive impairment | Day 1
  The level of cognitive impairment will be assessed by the cognitive score as per the Unified Huntington's Disease Rating Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Henri-Mondor, Créteil
  - Centre Hospitalier Universitaire de Bordeaux, Talence